

## STATISTICAL ANALYSIS PLAN

TITLE: Modulation of long-term memory by the experience of pain during sedation with anesthetics

NCT NUMBER: NCT02515890

PRINCIPAL INVESTIGATOR: Keith M. Vogt, M.D., Ph.D.

Dept. of Anesthesiology Montefiore Hospital, Suite 467

3459 Fifth Avenue, Pittsburgh, PA 15213

Telephone: 412-999-8570

**CO-INVESTIGATORS:** 

Julie Fiez, PhD James W. Ibinson, MD, PhD

Psychology & Neuroscience Anesthesiology

605 LRDC Montefiore Hospital, Suite 467

3939 O'Hara Street 3459 Fifth Avenue, Pittsburgh, PA 15213

Pittsburgh, PA 15260

SOURCE OF SUPPORT: Foundation for Anesthesia Education and Research

Department of Anesthesiology, UPMC



## Statistical Analysis Plan

TITLE: Modulation of long-term memory by the experience of pain during sedation with anesthetics

## **Primary Outcome: Memory Testing**

Explicit memory testing occurred the day following the drug administration and memory encoding session. Recognition testing was employed, using the well-known Remember-Know-New (RKN) scheme (Migo, Mayes et al. 2012). Recollection (for specific details) was indicated by a Remember response, while a Know response indicated familiarity. All words heard during the previous day were played intermixed with an equal number of foils, in randomized order. Memory performance was evaluated using d'. Statistical comparisons were performed in SPSS Statistics 23 (IBM, New York, NY) using a Bonferroni-corrected P < .05 as the threshold for significance.

The signal detection metric, d', was calculated with formula: z(hits) – z(false alarms), where z() refers to the cumulative Gaussian distribution function, hits are previously-heard items recognized, and false alarms are foils incorrectly recognized. The average d' score for performance in each drug condition (saline, midazolam, and ketamine) are calculated and compared.